CLINICAL TRIAL: NCT04301258
Title: ProChondrix® CR Articular Cartilage Restoration Evaluation (PACE) Registry
Status: Terminated | Type: Observational
Why Stopped: Duplicative data/insufficient enrollment
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Other Study IDs: REG-PRO-002
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cartilage Injury; Cartilage Damage
Keywords: Cartilage; Cartilage Injury; Cartilage Repair; Cartilage Damage; Cartilage Lesion; Cartilage Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Articular Cartilage Defect of the Knee: Patients, who undergo an articular cartilage repair of the knee using ProChondrix CR.
  Interventions: Other: Articular cartilage repair
- Articular Cartilage Defect of the Ankle: Patients, who undergo an articular cartilage repair of the ankle using ProChondrix CR.
  Interventions: Other: Articular cartilage repair
- Articular Cartilage Defect of the Foot: Patients, who undergo an articular cartilage repair of the foot using ProChondrix CR.
  Interventions: Other: Articular cartilage repair
- Articular Cartilage Defect of the Hip: Patients, who undergo an articular cartilage repair of the hip using ProChondrix CR.
  Interventions: Other: Articular cartilage repair

INTERVENTIONS:
Other: Articular cartilage repair — Patient reported outcomes will be collected on patients who have had a cartilage repair procedure using ProChondrix CR in the knee, hip, foot or ankle.
  Other Names: ProChondrix CR

SUMMARY:
The primary objective of this registry is to obtain long-term outcomes on ProChondrix CR in cartilage repair procedures of the knee, ankle, foot and hip.

DETAILED DESCRIPTION:
This multi-center, observational registry will be used to evaluate the effectiveness of ProChondrix CR in patients who undergo treatment for an articular cartilage defect in the knee, ankle, foot or hip.

This registry will be performed at up to 30 clinical sites across the United States.

Patient follow-up will occur following an articular cartilage repair procedure in which the patient receives ProChondrix CR. During this follow-up period, each patient will be evaluated at least four (4) times at: 3, 6, 12 and 24 months after surgical intervention and will continue annually for as long as patients are willing to fill out questionnaires and outcomes assessments up to 10 years post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by physician to have a cartilage defect in the knee, ankle, foot or hip that requires surgical intervention;
* Will be having, or has had, a cartilage repair procedure using ProChondrix CR;
* Has the ability to understand the requirements of the registry, to provide written informed consent and to comply with the registry protocol;

Exclusion Criteria:

• Is a ward of the state, prisoner, or transient.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients, who diagnosed by their treating physician, have a cartilage defect in the knee, ankle, foot or hip that requires surgical intervention utilizing ProChondrix CR.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Long-Term Outcomes of ProChondrix CR | 10 Years Post-Operative
  Obtain long-term results on patients who have undergone an articular cartilage repair procedure using ProChondrix CR, as assessed by patient reported outcomes.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Southern Alabama, Mobile, Alabama
  - Rocky Mountain Foot and Ankle Center, Wheat Ridge, Colorado
  - CAO Research Foundation, Washington D.C., District of Columbia
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Beacon Orthopaedics & Sports Medicine, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No